CLINICAL TRIAL: NCT00001695
Title: Survey of the Use of Alternative Medical Therapies in Adult Cancer Patients Enrolled in Phase I Clinical Trials
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 980098; 98-C-0098
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-01

CONDITIONS: Neoplasm
Keywords: Complementary Medicine; Unproven Treatments; Herbal
MeSH Terms: conditions — Neoplasms

SUMMARY:
Simultaneous use of alternative or complementary medical therapies by cancer patients undergoing conventional medical treatment is extremely common and may not always be disclosed to the patient's treating physician. Cancer patients undergoing Phase I therapy on clinical trials constitute a special population of patients, since by definition, their prescribed therapy is scientifically unproven in terms of efficacy. Phase I patients are closely monitored for adverse effects in order to identify and characterize the toxicities and to define a tolerable dose of their experimental treatment. Thus, the unrecognized use of alternative therapies by patients actively enrolled in phase I trials may potentially confound rational drug development by causing adverse side effects or by contributing to drug interactions. Examples of clinical toxicities induced by alternative medical treatments include liver dysfunction or renal failure caused by herbal preparations, or hematologic abnormalities, such as eosinophilia-myalgia syndrome caused by tryptophan food supplements. Therefore, it is important to document and determine the prevalence of alternative therapy use in this specific patient population; however, this issue has not previously been examined in a scientifically rigorous manner. We propose to conduct a survey and interview study of phase I cancer patients enrolled in ongoing clinical trials at the National Cancer Institute to determine the prevalence of alternative therapy use in this population. This study will also examine patient attitudes and perceptions regarding their use of alternative therapy as compared with their scientifically-sanctioned phase I experimental therapy. This information has important implications for drug development.

DETAILED DESCRIPTION:
Simultaneous use of alternative or complementary medical therapies by cancer patients undergoing conventional medical treatment is extremely common and may not always be disclosed to the patient's treating physician. Cancer patients undergoing Phase I therapy on clinical trials constitute a special population of patients, since by definition, their prescribed therapy is scientifically unproven in terms of efficacy. Phase I patients are closely monitored for adverse effects in order to identify and characterize the toxicities and to define a tolerable dose of their experimental treatment. Thus, the unrecognized use of alternative therapies by patients actively enrolled in phase I trials may potentially confound rational drug development by causing adverse side effects or by contributing to drug interactions. Examples of clinical toxicities induced by alternative medical treatments include liver dysfunction or renal failure caused by herbal preparations, or hematologic abnormalities, such as eosinophilia-myalgia syndrome caused by tryptophan food supplements. Therefore, it is important to document and determine the prevalence of alternative therapy use in this specific patient population; however, this issue has not previously been examined in a scientifically rigorous manner. We propose to conduct a survey and interview study of phase I cancer patients enrolled in ongoing clinical trials at the National Cancer Institute to determine the prevalence of alternative therapy use in this population. This study will also examine patient attitudes and perceptions regarding their use of alternative therapy as compared with their scientifically-sanctioned phase I experimental therapy. This information has important implications for drug development.

ELIGIBILITY:
Patients must be registered and actively participating in a Phase I clinical trial in the Division of Hematology/Oncology, National Naval Medical Center.

Patients must be able to give signed, informed consent.

Patients must be greater than or equal to 18 years old.

Patients must be medically well enough to be interviewed and to fill out the study questionnaire.

Patients must not have been previously enrolled in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 125
Dates: Start 1998-04; Study Completion 2002-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Eisenberg DM, Kessler RC, Foster C, Norlock FE, Calkins DR, Delbanco TL. Unconventional medicine in the United States. Prevalence, costs, and patterns of use. N Engl J Med. 1993 Jan 28;328(4):246-52. doi: 10.1056/NEJM199301283280406. PMID 8418405
- [Background] Cassileth BR, Chapman CC. Alternative and complementary cancer therapies. Cancer. 1996 Mar 15;77(6):1026-34. No abstract available. PMID 8635119